CLINICAL TRIAL: NCT04418934
Title: Clinical Investigation to Evaluate the Hemanext® Red Blood Cell Processing System for Extended Storage of Leukoreduced Red Blood Cells With CP2D Anticoagulant and AS-3 Additive - Pivotal Trial
Brief Title: Clinical Investigation to Evaluate the Hemanext® Red Blood Cell Processing System for Extended Storage of Leukoreduced Red Blood Cells
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Grant application for study was rejected
Sponsor: Hemanext (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CLIN-0004
Record Dates: First submitted 2020-05-26; First posted 2020-06-05 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Whole Blood Donations and Leukoreduction
Keywords: Red Blood Cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Investigational Product (Experimental): Blood product from these donors will be processed and stored using the Hemanext One device.
  Interventions: Device: Hemanext One
- Control Product (No Intervention): Blood product from these donors will be stored in a Haemonetics Leukotrap Whole Blood System.

INTERVENTIONS:
Device: Hemanext One — Leukoreduced red blood cell product from donors in the Investigational Product arm will be processed in the Hemanext Oxygen Reduction Bag for 3 hours and then transferred to the Hemanext Storage Bag and stored for 56 days at 1-6°C.
  Arms: Investigational Product

SUMMARY:
The primary goal of Hemanext Inc. is to improve the safety and efficacy of transfusion therapy through novel storage methods potentially improving their quality across the storage cycle. Based on our review of the pertinent literature, there is substantial evidence suggesting that prolonged exposure to oxygen during storage results in oxidative damage to the red blood cells (RBC) over the course of storage leading to decreased therapeutic potential. Therefore, removal of oxygen from red blood cell products prior to storage has potential to preserve the cells in a more physiologically relevant state and improve the clinical outcomes of patients that receive blood transfusions in a variety of therapeutic realms1.

Currently, Hemanext Inc. has focused on the design and development of a dual compartment bag system designated as the Hemanext Red Blood Cell Processing System (Hemanext). After standard processing of donated whole blood units into leukoreduced packed red blood cells (LR-RBCs) in AS-3 additive solution, the LR-RBCs would then be placed in the oxygen reduction bag (ORB) processing bag which allows for the rapid diffusion of oxygen out of the blood, through a sterile, oxygen-permeable membrane, and into iron-based oxygen sorbents. After processing, the blood is transferred again from the ORB into the Hemanext Storage Bag (HSB) which will preserve the hypoxic state of the LR-RBC product for the duration of cold storage.

The COVID-19 crisis has placed unprecedented pressure on the US blood supply security. The pandemic has caused blood supplies to fall precipitously, placing all transfusion recipients at acute risk. Hemanext has developed a technology over 12 years with support from 6 NIH grants and contracts that can substantially mitigate the damage done to the blood supply by this COVID-19 crisis and strengthen the ability of the US blood supply to withstand the effects of future crises. Limited shelf life is a key component in exacerbating the current blood supply crisis. Successful completion of this project will allow earliest possible availability (within 9-12 months) of the high quality Hemanext RBC with significantly extended shelf life. Even without shelf life extension, the higher quality Hemanext RBC showed a reduction of >50% of blood volume required for resuscitation from hemorrhage in a pre-clinical rodent model. Further enhancement of the quality of Hemanext RBC is expected to improve still further the efficacy of Hemanext blood and further to reduce the transfusion volume needed to achieve treatment objectives. In addition, extending the shelf life of the Hemanext RBC will provide greater inventory flexibility to avoid the devastating impact of major blood shortages due to reduced donor activity during threats to blood security such a COVID-19 pandemics and other crises.

ELIGIBILITY:
Inclusion Criteria:

Study donor must be ≥ 18 years of age. Study donor must be ≥ 110 pounds. Study donor's body temperature must be ≤ 37.5°C / 99.5°F (oral). Study donor's hemoglobin must be ≥12.5 g/dL if female and ≥13.0 g/dL if male. Study donor's hematocrit must be ≥ 38% if female and ≥39% if male.Study participants must meet EITHER hemoglobin or hematocrit criteria.

Study donor must meet all criteria per respective site's Research Blood Donation Record (BDR).

Study donor's most recent single RBC unit donation must have been ≥56 days prior to study donation.

Study donor's most recent double RBC unit donation must have been ≥ 112 days prior to study donation.

Study donor must have consented to study participation by reviewing and having expressed understanding the site-respective IRB-approved informed consent form prior to undergoing any study related procedures.

Study donor's testing results from collected blood does not indicate a risk of transfusion-transmitted disease (TTD)*.

Study donors must agree to report adverse events from the time of signing the informed consent to twenty-four hours following the end of their active study involvement.

Female study donors must not be pregnant, expected to be pregnant or breastfeeding.

Female donors who participate in the in vivo portion of the study:

Women of child-bearing age must not be pregnant as determined by a negative pregnancy test prior to each re-infusion. If acceptable by local procedures, post-menopausal or surgically sterile women may be exempt from the pregnancy testing requirement.

Exclusion Criteria:

Study donor is < 18 years of age. Study donor < 110 pounds. Study donor's body temperature is > 37.5°C / 99.5°F (oral). Study donor's hemoglobin is < 12.5 g/dL if female and < 13.0 g/dL if male. Study donor's hematocrit is < 38% if female and < 39% if male. Study donor does not meet all criteria per respective site's Research Blood Donation Record (BDR).

Study donor's most recent single RBC unit donation was < 56 days prior to study donation.

Study donor's most recent double RBC unit donation was < 112 days prior to study donation.

Study donor has not consented to study participation. Study donor's testing results from collected blood does indicate a risk of transfusion-transmitted disease (TTD)*.

Female donors who participate in the in vivo portion of the study: study donor is pregnant, expected to be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
% of Red Blood Cells With Hemolysis | Day 56 of storage
  Percentage of packed Red Blood Cell units with hemolysis at day 56 of storage.
Dual Label 24 Hour In Vivo % Recovery of Red Blood Cells | Day 56 of storage
  The mean 24-hour, post-transfusion, in vivo red blood cell recovery.
% Red Blood Cells Recovered Post-Filtration | Post-Filtration on Day 0
  Percentage of red blood cells recovered after the filtration process.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Cancelas, MD, PhD, Principal Investigator — Hoxworth Blood Center; Philip Howard, MD, Principal Investigator — American Red Cross Mid-Atlantic Research Facility
Locations (2):
- United States (2):
  - Hoxworth Blood Center, University of Cincinnati, Cincinnati, Ohio
  - American Red Cross Mid-Atlantic Research Facility, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No